CLINICAL TRIAL: NCT05143866
Title: Closing the Treatment Gap: A Pilot Study of Evidence-based Guided Self-Help for the Treatment of Binge Eating and Related Disordered Eating
Brief Title: A Pilot Study of Evidence-based Guided Self-help for the Treatment of Binge Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Eating Disorders Association (Other)
Responsible Party: Principal Investigator, Zafra Cooper, Professor of Psychiatry (adjunct), Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2000031521; No NIH funding (Other: 12.08.23)
Record Dates: First submitted 2021-11-16; First posted 2021-12-03 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Binge-Eating Disorder; Binge Eating
MeSH Terms: conditions — Binge-Eating Disorder; Bulimia

STUDY DESIGN:
Intervention Model Description: Feasibility with pre post assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-help CBT (Experimental): Evidence based book detailing self-help program to follow plus Telephone support from a non specialist guide
  Interventions: Behavioral: Cognitive behavioral therapy guided self help (CBTgsh)

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy guided self help (CBTgsh) — Based on evidence based cognitive behavioral treatment for eating disorders. Self-help version described in self-help book. Participant follows self-help program with encouragement and support of a non specialist guide

SUMMARY:
The purpose of the present pilot study is to evaluate the feasibility, acceptability and likely effectiveness of an evidence-based guided self-help intervention for binge eating and related disordered over-eating in those unable to access clinician provided treatments. If feasible, acceptable and likely to be effective, such interventions could be made available more widely as an early intervention to those in need. Such interventions have the potential to improve quality of life by removing or ameliorating symptoms that impair psychological and social functioning. Eligible participants will receive the guided self-help intervention - an evidence-based self help program in the form of a self-help book plus telephone support and encouragement to follow the program provided by specially trained help-line volunteers. Support completing the self-help program will be provided over a period of 4 months and participants will be followed up for a year after completion of the intervention. Participants will be asked to complete brief online assessments before starting the program, at the end of 4 months when they complete the program and at 6 month and 12 month follow up.

ELIGIBILITY:
Inclusion Criteria:

* Participant contacted National Eating Disorder Association (NEDA) with binge eating problems or disordered overeating
* Completed NEDA screen and study screen
* Age 18 and over
* Able to speak, understand and read English
* Consenting to guided self-help and completing study assessments

Exclusion Criteria:

* Currently receiving treatment for an eating disorder
* Self-reported weight body mass index (BMI) <20
* Reported self-induced vomiting, laxative or diuretic use (purging)
* Reports suicidal ideation
* Breast feeding or pregnant
* Receiving treatment for co-existing psychiatric condition (e.g., bipolar disorder, psychotic illness, drug or alcohol dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of providing intervention-consent | week 0 (baseline)
  Percentage of eligible participants who consent to intervention
Feasibility of providing intervention-completion Participants' ratings of satisfaction with the intervention | 16 weeks
  Percentage of eligible participants who complete intervention
Ratings of Acceptability of intervention to participants | At Baseline - before start of intervention
  Participants' ratings of suitability of intervention on visual analogue scale with anchors of strongly agree to strongly disagree
Ratings of Acceptability of intervention to participants | 16 weeks
  Participants' ratings of suitability of intervention on visual analogue scale with anchors strongly agree to strongly disagree
Ratings of Acceptability of intervention to participants | 10 months
  Participants' ratings of suitability of intervention on visual analogue scale with anchors strongly agree to strongly disagree
Ratings of Acceptability of intervention to participants | 16 months
  Participants' ratings of suitability of intervention on visual analogue scale with anchors strongly agree to strongly disagree
Ratings of participants' satisfaction with intervention with anchors strongly agree to strongly disagree | 16 weeks
  Participants rating of satisfaction with intervention on visual analogue scale with anchors strongly agree to strongly disagree
Ratings of participants' satisfaction with intervention | 10 months
  Participants rating of satisfaction with intervention on visual analogue scale with anchors strongly agree to strongly disagree
Ratings of participants' satisfaction with intervention | 16 months
  Participants rating of satisfaction with intervention on visual analogue scale with anchors strongly agree to strongly disagree

SECONDARY OUTCOMES:
Likely effectiveness -Eating difficulties | week 0 (baseline) and week 16 (end of intervention)
  Change in global score on a well validated self-report measure of eating disorder attitudes and behavior-Eating Disorder Questionnaire. Possible range from 0 - 6 where higher score indicates worse symptoms.
Likely effectiveness -Eating difficulties | week 0 (baseline) and week 64 (48 weeks/1 year after end of intervention)
  Change in global score on a well validated self-report measure of eating disorder attitudes and behavior-Eating Disorder Questionnaire. Possible range from 0 - 6 where higher score indicates worse symptoms.
Likely effectiveness - impairment due to eating difficulties | Week 0 (baseline) and week 16 (end of intervention)
  Change in impairment due to eating difficulties score on well validated self report measure the Clinical Impairment assessment (CIA). Possible scores range from 0 (no impairment ) to 48 (highest level of impairment).
Likely effectiveness - impairment due to eating difficulties | Week 0 (baseline) and week 64 (48 weeks/1 year after end of intervention)
  Change in impairment due to eating difficulties score on well validated self report measure the Clinical Impairment assessment (CIA). Possible scores range from 0 (no impairment ) to 48 (highest level of impairment).
Likely effectiveness - depression | Week 0 and week 16 (end of intervention)
  Change in depression scores on well validated self report measure, Patient Health Questionnaire (PHQ 9). Possible scores 0 (no depressed mood) to 27 (highest levels of depressive symptoms.
Likely effectiveness - depression | Week 0 and week 64 (48 weeks/1 Year after end of intervention)
  Change in depression scores on well validated self report measure, Patient Health Questionnaire (PHQ 9). Possible scores 0 (no depressed mood) to 27 (highest levels of depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Gabe Gavito, MS, Study Director — National Eating Disorders Association
Locations (1):
- Yale Medical School Department of Psychiatry, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No